CLINICAL TRIAL: NCT00158665
Title: A Comparison of One Versus Two Doses of Influenza Vaccine in Children Aged 5-8 Years of Age Receiving Influenza Vaccine for the First Time
Brief Title: A Comparison of One Versus Two Doses of Influenza Vaccine in Children 5-8 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC Protocol 4258; VSD contract #200-2002-00732 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Immunization; Flu; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving vaccine (Experimental): 2 0.5 ml doses of '04-05 Trivalent Influenza Vaccine 4 weeks apart.
  Interventions: Biological: 2 0.5 ml doses of '04-05 Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: 2 0.5 ml doses of '04-05 Trivalent Influenza Vaccine — 2 0.5 ml doses of '04-05 Trivalent Influenza Vaccine

SUMMARY:
The purpose of the study was to find out if children 5 through 8 years of age who are getting influenza vaccine for the first time should get one or two doses.

DETAILED DESCRIPTION:
Currently, two doses of influenza vaccine are recommended for children younger than 9 years receiving influenza vaccine for the first time. While the scientific support for 2 doses of vaccine in infants and toddlers is sound, the need for 2 doses of vaccine for adequate immunogenicity in older children is less certain. If the immunogenicity of a one-dose vaccine regimen is comparable to a two-dose regimen, then one dose would be preferable for reasons of safety, practicality and economics, and would reduce a major barrier to vaccination in this injection-adverse age group. This study compared the immunogenicity and reactogenicity of one versus two doses of influenza vaccine in children aged 5 to 8 years old receiving influenza vaccine for the first time. All children enrolled in the study received two doses of vaccine, and the immune response after one dose of vaccine was compared to the immune response after two doses of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent children who are at least 5 and no more than 8 years of age on the date of the first vaccination.
* Parents able to give informed consent and child available for all study visits.
* Family able to understand and comply with planned study procedures.
* Family must have telephone accessibility.

Exclusion Criteria:

* Previous receipt of influenza vaccine of any kind (shot or nasal spray).
* Active cancer or blood system abnormalities such as leukemia.
* Immunocompromising illnesses or current receipt of immunosuppressive agents
* Allergy to eggs or egg protein, or to gentamicin (an antibiotic that is present in trace amounts in the vaccine).
* Any acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses.

Temporary Exclusion Criteria:

Acute disease, defined as the presence of moderate or severe illness with or without fever, at the time of enrollment. Influenza vaccine may be administered to children with minor illnesses, such as diarrhea, mild upper respiratory infection and low-grade febrile illness with an oral temperature <100.4 F.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2004-08; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Comparison of antibody response after 1 dose of influenza vaccine with that after 2 doses of influenza vaccine. | Blood samples were obtained at 3 time points, before dose 1 of vaccine, 4 weeks after receipt of dose 1 and before dose 2, and 4 weeks after dose 2 of vaccine.

SECONDARY OUTCOMES:
To describe and compare the safety profile after 1 and 2 doses of vaccine. | Study diaries were kept from the day of vaccination daily for the 4 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Jackson, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Result] Neuzil KM, Jackson LA, Nelson J, Klimov A, Cox N, Bridges CB, Dunn J, DeStefano F, Shay D. Immunogenicity and reactogenicity of 1 versus 2 doses of trivalent inactivated influenza vaccine in vaccine-naive 5-8-year-old children. J Infect Dis. 2006 Oct 15;194(8):1032-9. doi: 10.1086/507309. Epub 2006 Sep 11. PMID 16991077